CLINICAL TRIAL: NCT02643485
Title: Dynamic Pedobarography With a New Insole After Forefoot Reconstruction
Brief Title: Pedobarographic Changes After Forefoot Reconstruction
Acronym: PEDfore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Harrasser, Dr., Technical University of Munich
Other Study IDs: 10111
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Plantar Foot Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Patients undergoing forefoot reconstruction of hallux valgus or hallux rigidus
  Interventions: Procedure: Forefoot surgery
- Control group: Healthy volunteers (Students)

INTERVENTIONS:
Procedure: Forefoot surgery — Forefoot surgery (Chevron, Scarf, Lapidus, Arthrodesis)
  Groups: Study group

SUMMARY:
Static pedobarography is routinely used for pre- and postoperative questions regarding plantar foot pressure. This Investigation does insufficiently detect dynamic Forces. Hence, dynamic pedobarography might give some important insights in detecting plantar foot pressure after forefoot reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Forefoot surgery for hallux valgus or rigidus planned at out departement

Exclusion Criteria:

* No given consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients planned for forefoot surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
AOFAS-Score (American Orthopedic Foot and Ankle Society) | 2 years

SECONDARY OUTCOMES:
Plantar Peak Pressure | 2 years
  Measuring will be performed by insole (Fa. Meticon) capable to detect plantar pressure in 80 regions of the sole of the foot

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger Eisenhart-Rothe, Prof., Study Director — Head of Orthopedic Dept.
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No